CLINICAL TRIAL: NCT02388724
Title: A Randomized, Double-Blind, Double-Dummy Phase 3 Study to Evaluate the Efficacy and Safety of Oral Once-Daily Administration of TAK-438 20 mg Compared to Lansoprazole 30 mg in the Treatment of Subjects With Erosive Esophagitis
Brief Title: Efficacy and Safety of Oral Once-Daily Vonoprazan (TAK-438) in Participants With Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-438_303; U1111-1138-4788 (Registry Identifier: UTN (WHO)); CTR20150040 (Registry Identifier: CNDA CTR)
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Erosive Esophagitis
Keywords: Drug therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vonoprazan 20 mg (Experimental): Vonoprazan 20 mg, tablet, orally, once daily and lansoprazole placebo-matching capsule, orally, once daily for up to 8 weeks.
  Interventions: Drug: Vonoprazan; Drug: Lansoprazole Placebo
- Lansoprazole 30 mg (Active Comparator): Lansoprazole 30 mg, capsule, orally, once daily and vonoprazan placebo-matching tablet, orally, once daily for up to 8 weeks.
  Interventions: Drug: Lansoprazole; Drug: Vonoprazan Placebo

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan tablets
  Other Names: TAK-438
  Arms: Vonoprazan 20 mg
Drug: Lansoprazole — Lansoprazole capsules
  Other Names: Prevacid
  Arms: Lansoprazole 30 mg
Drug: Vonoprazan Placebo — Vonoprazan placebo-matching tablets
  Arms: Lansoprazole 30 mg
Drug: Lansoprazole Placebo — Lansoprazole placebo-matching capsules
  Arms: Vonoprazan 20 mg

SUMMARY:
The purpose of the study is to demonstrate the efficacy of vonoprazan (TAK-438) versus lansoprazole in the treatment of erosive esophagitis classified as Los Angeles (LA) classification grades A to D at Week 8.

DETAILED DESCRIPTION:
The drug being tested in this study is called vonoprazan. Vonoprazan is being tested to treat people who have erosive esophagitis. This study will look at mucosal healing of people who take vonoprazan versus lansoprazole.

This study will enroll approximately 480 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Vonoprazan 20 mg
* Lansoprazole 30 mg

All participants will be asked to take one tablet and one capsule at the same time each day throughout the study. All participants will be asked to record daytime and nighttime (during sleep) subjective symptoms in a diary on a daily basis.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is up to 11 weeks. Participants will make multiple visits to the clinic, and will be contacted by telephone 7-14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Has been confirmed in an endoscopy to have erosive esophagitis, ie, the Los Angeles (LA) classification grades A to D within 7 days of the start of the Day 1 (Visit 2).

   Note: The recruitment goal is to ensure that those with LA classification grade C/D will account for more than 30% of all participants enrolled (144/480), with no further recruitment of those with grade A/B considered when they account for more than 70% (336/480) of all participants.
4. Is aged 18 years old or older (or the local age of consent if that is older), male or female, at the time of signing an informed consent, and is being treated on an outpatient basis for erosive esophagitis, including those admitted temporarily for examination.
5. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study.

Exclusion Criteria:

1. Has received any investigational compound within 84 days prior to the start of the Observation phase.
2. Has received TAK-438 in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has, in the judgment of the investigator, clinically significant abnormal hematological parameters of hemoglobin, hematocrit, or erythrocytes at Screening.
5. Has a history or clinical manifestations of serious central nerve system (CNS), cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urological, endocrine or hematological disease.
6. Has a history of hypersensitivity or allergies to TAK-438 (including its excipients*) or to proton pump inhibitors (PPIs).

   *D-mannitol, crystalline cellulose, hydroxypropyl cellulose, fumaric acid, croscarmellose sodium, magnesium stearate, hypromellose, macrogol 6000, titanium oxide, yellow iron sesquioxide and iron sesquioxide.
7. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Observation Phase (Visit 1).
8. Is required to take excluded medications.
9. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
10. Has participated in another clinical study within the past 30 days from Visit 1.
11. Has co-morbidities that could affect the esophagus (eosinophilic esophagitis, esophageal varices, scleroderma, viral or fungal infection, esophageal strictures), a history of radiotherapy or cryotherapy for the esophagus; those with corrosive or physiochemical injury (with the possible inclusion in the study of those with Schatzki's ring or Barrett's esophagus).
12. Has a history of surgical procedures that may affect the esophagus (eg, fundoplication and mechanical dilatation for esophageal strictures excluding Schatzki's ring) or a history of gastric or duodenal surgery excluding endoscopic removal of benign polyps.
13. Developed acute upper gastrointestinal bleeding, gastric ulcer (a mucosal defect with white coating) or duodenal ulcer (a mucosal defect with white coating), within 30 days before the start of the Observation Phase (Visit 1) (with the possible inclusion of those with gastric or duodenal erosion).
14. Has Zollinger-Ellison syndrome or gastric acid hypersecretion or a history of gastric acid hypersecretion.
15. Is scheduled for surgery that requires hospitalization or requires surgical treatment during his/her participation in the study.
16. Has a history of malignancy or was treated for malignancy within 5 years before the start of the Observation Phase (Visit 1) (the participant may be included in the study if he/she has cured cutaneous basal cell carcinoma or cervical carcinoma in situ).
17. Has acquired immunodeficiency syndrome (AIDS) or hepatitis, including hepatitis virus carriers: hepatitis B surface antigen (HBsAg) positive, or hepatitis C virus (HCV)-antibody-positive (the participant may be included in the study if he/she is HCV-antigen or HCV-ribonucleic acid [RNA]-negative).
18. Laboratory tests performed at the start of the Early Observation Phase (visit 1) revealed any of the following abnormalities in the participant:

    1. Creatinine levels: >2 mg/dL (>177 μmol/L).
    2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST), or total bilirubin levels: > upper limit of normal (ULN).
19. Is active in the Screening Period after the closure of enrollment identified by the Sponsor or the number of participants randomized with LA classification A/B or C/D have reached the required sample size.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (64):
- China (32):
  - Beijing Chao Yang Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical Univeristy, Beijing, Beijing Municipality
  - PLA.The Military General Hospital of Beijing, Beijing, Beijing Municipality
  - Fuzhou General Hospital of Nanjing Military Command, Fuzhou, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The 2nd Xiangya Hospital Central South University, Changsha, Hu'nan
  - Chenzhou No.1 People's Hospital, Chenzhou, Hu'nan
  - Union Hospital of Tongji Medical College of Huazhong Science and Techology University, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Techology, Wuhan, Hubei
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Province People's Hospital, Nanjing, Jiangsu
  - No.2 Hospital Affiliated to Jilin University, Changchun, Jilin
  - Jilin central Hospital, Jilin, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia Hui
  - Ruijin Hospital, Shanghai Jiaotong Uni. School of Med., Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - TongJi Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The 2nd Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The First Affiated Hospital of Kunming Medical College, Kunming, Yun'nan
  - 2nd Affiliated Hospital, Zhejiang Univ. School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - 1st Affiliated Hospital of Zhejiang University, Hangzhou
  - The First Affiliated Hospital of NanChang University, Nanchang
  - The Affiliated DrumTower Hospital of Nanjing University, Nanjing
  - Tianjin
- Malaysia (8):
  - Hospital Sultana Bahiyah, Alor Star, Kedah
  - Hospital Universiti Sains Malaysia, Kelantan, Kelantan
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Queen Elizabeth, Kota Kinabalu, Sabah
  - Hospital Ampang, Ampang, Selangor
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
- South Korea (12):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Gyeonggi-do
  - Kyungpook National University Medical Center, Daegu, Gyeongsangbuk-do
  - Wonkwang University School Of Medicine & Hospital, Iksan-si, Jeollabuk-do
  - Pusan National University Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Marys Hospital, Seoul
- Taiwan (12):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - Cheng Ching General Hospital-Chung Kang Branch, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan

REFERENCES:
- [Derived] Xiao Y, Zhang S, Dai N, Fei G, Goh KL, Chun HJ, Sheu BS, Chong CF, Funao N, Zhou W, Chen M. Phase III, randomised, double-blind, multicentre study to evaluate the efficacy and safety of vonoprazan compared with lansoprazole in Asian patients with erosive oesophagitis. Gut. 2020 Feb;69(2):224-230. doi: 10.1136/gutjnl-2019-318365. Epub 2019 Aug 13. PMID 31409606

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 56 investigative sites in China, Korea, Taiwan, and Malaysia from 24 March 2015 to 27 July 2017.
Pre-assignment Details: Participants with a diagnosis of erosive esophagitis were enrolled in a 1:1 ratio in one of two treatment groups, TAK-438 20 mg once daily (QD) or lansoprazole 30 mg QD.
Period: Overall Study
Arm/Group | Vonoprazan 20 mg | Lansoprazole 30 mg
Started | 244 | 237
Safety Set: Randomized But Not Treated | 0 | 2
Completed (Completed=Completed Treatment) | 232 | 224
Not Completed | 12 | 13
Not completed — Reason not Specified | 0 | 1
Not completed — Major Protocol Deviation | 3 | 3
Not completed — Pretreatment Event/Adverse Event | 3 | 2
Not completed — Voluntary Withdrawal | 6 | 5
Not completed — Randomized but not Treated | 0 | 2

BASELINE CHARACTERISTICS:
Population: Randomized set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vonoprazan 20 mg | Lansoprazole 30 mg | Total
Number analyzed (Participants) | 244 | 237 | 481
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (13.16) | 53.8 (12.53) | 53.9 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 58 | 126
  Male | 176 | 179 | 355
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 244 | 237 | 481
Region of Enrollment [Count of Participants; unit: Participants]
  Asia: China | 143 | 133 | 276
  Asia: Malaysia | 21 | 24 | 45
  Asia: South Korea | 52 | 55 | 107
  Asia: Taiwan | 28 | 25 | 53
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 166.1 (8.24) | 166.3 (8.80) | 166.2 (8.52)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] — Population: Data for 2 participants in the Lansoprazole 30 mg arm were missing because they were randomized, but terminated early due to voluntary withdrawal.
  kilograms (kg)
    number analyzed (Participants) | 244 | 235 | 479
    (all) | 68.48 (12.311) | 70.26 (12.133) | 69.35 (12.243)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Population: Data for 2 participants in the Lansoprazole 30 mg arm were missing because they were randomized, but terminated early due to voluntary withdrawal.
  kilograms per square meter (kg/m^2)
    number analyzed (Participants) | 244 | 235 | 479
    (all) | 24.70 (3.389) | 25.31 (3.430) | 25.00 (3.419)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 157 | 137 | 294
  Current Smoker | 48 | 64 | 112
  Ex-Smoker | 39 | 36 | 75
Consumption of Alcohol [Count of Participants; unit: Participants]
  Drink Everyday | 13 | 12 | 25
  Drink a Couple of Days Per Week | 32 | 40 | 72
  Drink a Couple of Days Per Month | 57 | 48 | 105
  Never Drink | 142 | 137 | 279
Consumption of Caffeine [Count of Participants; unit: Participants] — Population: The number of participants in the Vonoprazan 20 mg arm with non-missing data obtained from the case report form / electronic data capture was 243.
  Participants
    Yes: number analyzed (Participants) | 243 | 237 | 480
    Yes | 58 | 52 | 110
    No: number analyzed (Participants) | 243 | 237 | 480
    No | 185 | 185 | 370
History of H. pylori Eradication Therapy [Count of Participants; unit: Participants]
  Yes (End of Treatment: Within the Past 1 Year) | 6 | 4 | 10
  Yes (End of Treatment: More than 1 Year) | 18 | 22 | 40
  No | 220 | 211 | 431
H. pylori Infection Status [Count of Participants; unit: Participants] — Population: The number of participants in the Vonoprazan 20 mg and Lansoprazole 30 mg arms with non-missing data obtained from the case report form / electronic data capture was 241 and 234, respectively.
  Participants
    Positive: number analyzed (Participants) | 241 | 234 | 475
    Positive | 36 | 38 | 74
    Negative: number analyzed (Participants) | 241 | 234 | 475
    Negative | 205 | 196 | 401
LA Classification for Diagnosis and Grading of Erosive Esophagitis [Count of Participants; unit: Participants] — Grade O (no mucosal breaks); Grade A (one or more mucosal breaks no longer than 5 millimeters [mm], none of which extends between the tops of the mucosal folds); Grade B (one or more mucosal breaks more than 5 mm long, none of which extends between the tops of 2 mucosal folds); Grade C (mucosal breaks that extend between the tops of 2 or more mucosal folds, but which involve less than 75% of esophageal circumference), Grade D mucosal breaks which involve at least 75% of esophageal circumference. Population: Data for 2 participants in the Lansoprazole 30 mg arm were missing because they were randomized, but terminated early due to voluntary withdrawal.
  Participants
    Grade O: number analyzed (Participants) | 244 | 235 | 479
    Grade O | 0 | 0 | 0
    Grade A: number analyzed (Participants) | 244 | 235 | 479
    Grade A | 76 | 83 | 159
    Grade B: number analyzed (Participants) | 244 | 235 | 479
    Grade B | 92 | 84 | 176
    Grade C: number analyzed (Participants) | 244 | 235 | 479
    Grade C | 58 | 58 | 116
    Grade D: number analyzed (Participants) | 244 | 235 | 479
    Grade D | 18 | 10 | 28
Barrett's Mucosa [Count of Participants; unit: Participants] — Population: Data for 2 participants in the Lansoprazole 30 mg arm were missing because they were randomized, but terminated early due to voluntary withdrawal.
  Participants
    Present (3 cm or Greater): number analyzed (Participants) | 244 | 235 | 479
    Present (3 cm or Greater) | 7 | 7 | 14
    Present (Less than 3 cm): number analyzed (Participants) | 244 | 235 | 479
    Present (Less than 3 cm) | 15 | 10 | 25
    Absent: number analyzed (Participants) | 244 | 235 | 479
    Absent | 216 | 212 | 428
    Unknown: number analyzed (Participants) | 244 | 235 | 479
    Unknown | 6 | 6 | 12
Esophageal Hiatal Hernia [Count of Participants; unit: Participants] — Population: Data for 2 participants in the Lansoprazole 30 mg arm were missing because they were randomized, but terminated early due to voluntary withdrawal.
  Participants
    Present (2 cm or Greater): number analyzed (Participants) | 244 | 235 | 479
    Present (2 cm or Greater) | 36 | 39 | 75
    Present (Less than 2 cm): number analyzed (Participants) | 244 | 235 | 479
    Present (Less than 2 cm) | 24 | 24 | 48
    Absent: number analyzed (Participants) | 244 | 235 | 479
    Absent | 180 | 166 | 346
    Unknown: number analyzed (Participants) | 244 | 235 | 479
    Unknown | 4 | 6 | 10
Diary for Gastrointestinal Symptoms: Mean Severity of Heartburn Symptoms [Mean (Standard Deviation); unit: score on a scale] — 0=None (no symptoms), 1=Mild (occasional symptoms, can be ignored, does not influence daily routine), 2=Moderate (symptoms cannot be ignored and/or occasionally influence daily routine), 3=Severe (symptoms present most of the day and/or regularly influence daily routine) Population: Data for 2 participants in the Lansoprazole 30 mg arm were missing because they were randomized, but terminated early due to voluntary withdrawal.
  score on a scale
    number analyzed (Participants) | 244 | 235 | 479
    (all) | 0.797 (0.7153) | 0.767 (0.6408) | 0.782 (0.6792)
Mean Severity of Gastric Acid Regurgitation [Mean (Standard Deviation); unit: score on a scale] — 0=None (no symptoms), 1=Mild (occasional symptoms, can be ignored, does not influence daily routine), 2=Moderate (symptoms cannot be ignored and/or occasionally influence daily routine), 3=Severe (symptoms present most of the day and/or regularly influence daily routine) Population: Data for 2 participants in the Lansoprazole 30 mg arm were missing because they were randomized, but terminated early due to voluntary withdrawal.
  score on a scale
    number analyzed (Participants) | 244 | 235 | 479
    (all) | 0.772 (0.6765) | 0.727 (0.6731) | 0.750 (0.6745)
Health-Related Quality of Life (HRQoL) EQ-5D-5L Index Value [Mean (Standard Deviation); unit: score on a scale] — The EQ-5D-5L Index assesses 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 response levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are combined and converted to a single index score. The lowest possible score is -0.39 (unable to walk, care for oneself, do usual activities; having extreme pain or discomfort; extreme anxiety or depression) and the highest is 1.00 (no problems in all 5 dimensions). Population: Data for 2 participants in the Lansoprazole 30 mg arm were missing because they were randomized, but terminated early due to voluntary withdrawal.
  score on a scale
    number analyzed (Participants) | 244 | 235 | 479
    (all) | 0.9503 (0.07278) | 0.9486 (0.06466) | 0.9495 (0.06885)
EuroQol-visual analogue scales (EQ VAS) Score [Mean (Standard Deviation); unit: score on a scale] — The EQ VAS is a questionnaire asking the participant to mark health status on a 20 cm vertical scale, ranging from 0 (worst health you can imagine) to 100 (best health you can imagine). Population: Data for 2 participants in the Lansoprazole 30 mg arm were missing because they were randomized, but terminated early due to voluntary withdrawal.
  score on a scale
    number analyzed (Participants) | 244 | 235 | 479
    (all) | 85.7 (10.88) | 85.2 (11.56) | 85.4 (11.21)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Endoscopic Healing of Erosive Esophagitis During the 8-Week Treatment Phase
Description: Endoscopic healing is defined as participants endoscopically diagnosed as Los Angeles classification grade O during the treatment phase. Grade O indicates there are no mucosal breaks in the mucosa.
Time Frame: 8 weeks
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline endoscopy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vonoprazan 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 238 | 230
percentage of participants | 92.4 [88.310 to 95.456] | 91.3 [86.890 to 94.607]
Statistical Analysis 1: Comparison: Vonoprazan 20 mg vs Lansoprazole 30 mg; Test type: Non-Inferiority — If the lower bound of the 95% confidence intervals of the difference was more than -10% (non-inferiority margin), non-inferiority for Vonoprazan relative to Lansoprazole was declared; Difference in percentages = 1.1, 95% CI 2-sided [-3.822 to 6.087]

2. Secondary Outcome: Percentage of Participants With Endoscopic Healing of Erosive Esophagitis After 2 Weeks and 4 Weeks of Treatment
Description: as for outcome 1
Time Frame: Week 2 and Week 4
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline endoscopy. Number analyzed is the number of participants with data available at the given time-point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vonoprazan 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 238 | 230
percentage of participants
  2 Weeks: number analyzed (Participants) | 236 | 227
  2 Weeks | 75.0 [68.970 to 80.391] | 67.8 [61.341 to 73.869]
  4 Weeks | 85.3 [80.146 to 89.538] | 83.5 [78.035 to 88.035]
Statistical Analysis 1: Comparison: Vonoprazan 20 mg vs Lansoprazole 30 mg; 2 Weeks; Test type: Superiority; Difference in percentages = 7.2, 95% CI 2-sided [-1.054 to 15.371]
Statistical Analysis 2: Comparison: Vonoprazan 20 mg vs Lansoprazole 30 mg; 4 Weeks; Test type: Superiority; Difference in percentages = 1.8, 95% CI 2-sided [-4.763 to 8.395]

3. Secondary Outcome: Number of Participants Reporting Who Had One or More Treatment-emergent Adverse Event (TEAE)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the drug.
Time Frame: On or after the start of study drug (Day 1) to 14 days after the last dose of study medication (up to 10 weeks)
Population: The safety analysis set (SAF) included all participants who took at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 244 | 235
Participants | 93 | 86

4. Secondary Outcome: Number of Participants With Markedly Abnormal Clinical Laboratory Findings
Description: Clinical Laboratory Safety tests included Chemistry, Hematology and Urinalysis. Number of participants with any markedly abnormal values in laboratory tests collected throughout study is reported. ALT = alanine aminotransferase, AST = aspartate aminotransferase, GGT = gamma-glutamyl transferase, CPK = creatine phosphokinase, BUN = blood urea nitrogen, LLN = lower limit of normal or lower reference limit, ULN = upper limit of normal or upper reference limit, g/L = grams per liter, U/L = units per liter, mmol/L = millimoles per liter, pmol/L = picomoles per liter.
Time Frame: From Day 1 to 14 days after the last dose of study medication (up to 10 weeks)
Population: The safety analysis set (SAF) included all participants who took at least 1 dose of study medication. The number analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 244 | 235
Participants
  Hemoglobin (<0.8 x LLN g/L): number analyzed (Participants) | 239 | 231
  Hemoglobin (<0.8 x LLN g/L) | 0 | 1
  Neutrophils (<0.5 x LLN %): number analyzed (Participants) | 239 | 230
  Neutrophils (<0.5 x LLN %) | 0 | 2
  Eosinophils (>2 x ULN %): number analyzed (Participants) | 239 | 230
  Eosinophils (>2 x ULN %) | 1 | 0
  Lymphocytes (>1.5 x ULN %): number analyzed (Participants) | 239 | 230
  Lymphocytes (>1.5 x ULN %) | 0 | 2
  ALT (>3 x ULN U/L): number analyzed (Participants) | 238 | 231
  ALT (>3 x ULN U/L) | 0 | 2
  AST (>3 x ULN U/L): number analyzed (Participants) | 238 | 231
  AST (>3 x ULN U/L) | 0 | 1
  GGT (>3 x ULN U/L): number analyzed (Participants) | 238 | 231
  GGT (>3 x ULN U/L) | 4 | 3
  CPK (>5 x ULN U/L): number analyzed (Participants) | 238 | 231
  CPK (>5 x ULN U/L) | 1 | 2
  Total Protein (>1.2 x ULN g/L): number analyzed (Participants) | 238 | 231
  Total Protein (>1.2 x ULN g/L) | 0 | 1
  BUN (>10.7 mmol/L): number analyzed (Participants) | 238 | 231
  BUN (>10.7 mmol/L) | 1 | 1
  Total Cholesterol (>7.72 mmol/L): number analyzed (Participants) | 238 | 231
  Total Cholesterol (>7.72 mmol/L) | 3 | 2
  Triglycerides (>2.5 x ULN mmol/L): number analyzed (Participants) | 238 | 231
  Triglycerides (>2.5 x ULN mmol/L) | 6 | 3
  Vitamin B12 (<92 pmol/L): number analyzed (Participants) | 236 | 227
  Vitamin B12 (<92 pmol/L) | 0 | 1

5. Secondary Outcome: Number of Participants With Markedly Abnormal Electrocardiogram (ECG) Findings
Description: Number of participants with any markedly abnormal 12-lead ECG findings is reported. bpm = beats per minute, msec = milliseconds, CHG= change from baseline.
Time Frame: From Day 1 to 14 days after the last dose of study medication (up to 10 weeks)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 244 | 235
Participants
  Heart Rate (<50 bpm): number analyzed (Participants) | 236 | 228
  Heart Rate (<50 bpm) | 6 | 7
  QT Interval (≥460 msec): number analyzed (Participants) | 236 | 228
  QT Interval (≥460 msec) | 7 | 10
  QTcF Interval (≥500, or ≥450 with CHG ≥30 msec): number analyzed (Participants) | 236 | 228
  QTcF Interval (≥500, or ≥450 with CHG ≥30 msec) | 3 | 5

6. Secondary Outcome: Number of Participants With Markedly Abnormal Vital Sign Measurements
Description: Number of participants with any markedly abnormal vital signs measurements is reported. Vital signs included body temperature (oral, tympanic, or infra-axillary measurement), sitting blood pressure (5 minutes), and pulse. °C = degrees Celsius, mmHg = millimeters of mercury, bpm = beats per minute.
Time Frame: From Day 1 to 14 days after the last dose of study medication (up to 10 weeks)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 244 | 235
Participants
  Body Temperature (<35.6 °C): number analyzed (Participants) | 241 | 231
  Body Temperature (<35.6 °C) | 10 | 3
  Body Temperature (>37.7 °C): number analyzed (Participants) | 241 | 231
  Body Temperature (>37.7 °C) | 2 | 0
  Systolic Blood Pressure (<85 mmHg): number analyzed (Participants) | 241 | 231
  Systolic Blood Pressure (<85 mmHg) | 1 | 1
  Diastolic Blood Pressure (>110 mmHg): number analyzed (Participants) | 241 | 231
  Diastolic Blood Pressure (>110 mmHg) | 1 | 0
  Pulse (<50 bpm): number analyzed (Participants) | 241 | 231
  Pulse (<50 bpm) | 2 | 2

7. Secondary Outcome: Change From Baseline in Serum Gastrin
Description: The change between the serum gastrin values collected at Weeks 2, 4, and 8 relative to baseline.
Time Frame: Baseline and Weeks 2, 4, and 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Vonoprazan 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 244 | 235
pmol/L
  Baseline: number analyzed (Participants) | 230 | 229
  Baseline | 2.77 (4.084) | 3.65 (8.622)
  Change at Week 2: number analyzed (Participants) | 220 | 219
  Change at Week 2 | 31.45 (28.995) | 8.33 (10.190)
  Change at Week 4: number analyzed (Participants) | 57 | 71
  Change at Week 4 | 29.68 (29.189) | 6.81 (9.969)
  Change at Week 8: number analyzed (Participants) | 30 | 31
  Change at Week 8 | 36.53 (37.108) | 4.71 (7.727)

8. Secondary Outcome: Change From Baseline in Serum Pepsinogen I
Description: The change between the serum pepsinogen I values collected at Weeks 2, 4, and 8 relative to baseline.
Time Frame: Baseline and Weeks 2, 4, and 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micrograms per liter (ug/L)
Arm/Group | Vonoprazan 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 244 | 235
micrograms per liter (ug/L)
  Baseline: number analyzed (Participants) | 238 | 231
  Baseline | 97.6 (53.54) | 99.8 (61.99)
  Change at Week 2: number analyzed (Participants) | 227 | 223
  Change at Week 2 | 456.5 (308.22) | 129.3 (138.24)
  Change at Week 4: number analyzed (Participants) | 57 | 71
  Change at Week 4 | 421.8 (324.06) | 118.3 (113.24)
  Change at Week 8: number analyzed (Participants) | 30 | 30
  Change at Week 8 | 326.8 (233.80) | 117.8 (98.03)

9. Secondary Outcome: Change From Baseline in Serum Pepsinogen II
Description: The change between the serum pepsinogen II values collected at Weeks 2, 4, and 8 relative to baseline.
Time Frame: Baseline and Weeks 2, 4, and 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Vonoprazan 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 244 | 235
ug/L
  Baseline: number analyzed (Participants) | 235 | 231
  Baseline | 7.5 (5.50) | 7.8 (5.77)
  Change at Week 2: number analyzed (Participants) | 227 | 225
  Change at Week 2 | 44.9 (31.31) | 8.8 (9.63)
  Change at Week 4: number analyzed (Participants) | 56 | 71
  Change at Week 4 | 40.7 (26.10) | 7.2 (5.99)
  Change at Week 8: number analyzed (Participants) | 29 | 31
  Change at Week 8 | 31.0 (20.03) | 8.0 (8.46)

ADVERSE EVENTS:
Time Frame: Up to 10 weeks (8 weeks of treatment and 2 weeks of post-treatment follow-up period)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal physical examination and laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Vonoprazan 20 mg | Lansoprazole 30 mg
All-Cause Mortality (participants affected / at risk) | 0/244 | 0/235
Serious Adverse Events (participants affected / at risk) | 3/244 | 3/235
Other Adverse Events (participants affected / at risk) | 13/244 | 4/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 20 mg (N=244) | Lansoprazole 30 mg (N=235)
Glaucoma (Eye disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 20 mg (N=244) | Lansoprazole 30 mg (N=235)
Blood gastrin increased (Investigations) | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study-related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT02388724/SAP_000.pdf
  • Study Protocol (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT02388724/Prot_001.pdf